CLINICAL TRIAL: NCT07346677
Title: Comparing of Sesame Oil, Nitroglycerin Ointment, and Aloe Vera Gel on Prevention of Phlebitis Induced by Chemotherapy
Brief Title: Comparing of Sesame Oil, Nitroglycerin Ointment, and Aloe Vera Gel
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Basrah (Other)
Collaborators: University of Baghdad (Other)
Responsible Party: Principal Investigator, Ali Malik Tiryag, Principle Investigator, University of Basrah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Prevention of Phlebitis
Record Dates: First submitted 2025-12-06; First posted 2026-01-16 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Chemotherapy
Keywords: sesame oil; aloe Vera gel; nitroglycerin ointment; phlebitis
MeSH Terms: conditions — Neoplasms; Phlebitis | interventions — Sesame Oil; Aloe vera gel; Green Or

STUDY DESIGN:
Intervention Model Description: True experimental design (comparative) this type of design allows the researcher to understand the best cause-and-effect relationship between independent variables (sesame oil, aloe Vera gel , nitroglycerin ointment) and dependent variables (phlebitis), among patient receiving chemotherapy(antimetabolites 5- fluorouracil , alkylating agents Cisplatin) and which intervention is more effective
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- sesame oil (Experimental): Sesame oil application is advised as a standard hospital treatment for patients receiving chemotherapy. It is possible to conduct a similar study with a large probability sample and in a variety of settings, allowing for greater generalization of the findings. The researchers will be applied 10 drops (3 mL) of 100% pure sesame oil in a circular motion for 5 minutes within 10 cm on the anterior forearm of the chemotherapy patient. They then gradually spread the oil around 10 cm toward the arm of the study group to improve absorption. Each 12 hours wasapplied 2-time morning and night. Record the frequency of phlebitis in the 24 and 48 hours after the intervention.
  Interventions: Biological: Sesame Oil
- Aloe Vera gel (Experimental): The researcher will soak the skin in 5 cc of Aloe vera gel, drawn with a syringe, in a circular motion for 20 minutes within 10 cm on the anterior forearm of the chemotherapy patient. They then gradually spread the gel around 10 cm toward the arm of the study group to improve absorption. Each 12 hours, 2 time morning and night, record the frequency of phlebitis in the 24 hours after the intervention.
  Interventions: Biological: Aloe vera gel
- nitroglycerin ointment (Experimental): The researchers will apply nitroglycerin ointment in a circular motion for 5 minutes over a 10 cm area on the anterior forearm of the chemotherapy patient. They then gradually spread the oil around 10 cm toward the arm of the study group to improve absorption. Each 12 hours, a 2-time morning and night record the frequency of phlebitis in the 24 and 48 hours after the intervention.
  Interventions: Biological: nitroglycerin ointment
- control (Other): without any intervention
  Interventions: Other: Control

INTERVENTIONS:
Biological: Sesame Oil — 10 drops (3 mL) of 100% pure sesame oil in a circular motion for 5 minutes within 10 cm on the anterior forearm of the chemotherapy patient. T
  Other Names: Yellow
  Arms: sesame oil
Biological: Aloe vera gel — soak the skin in 5 cc of Aloe vera gel, drawn with a syringe, in a circular motion for 20 minutes within 10 cm on the anterior forearm of the chemotherapy patient.
  Other Names: green
  Arms: Aloe Vera gel
Other: Control — without any intervention
  Other Names: white
  Arms: control
Biological: nitroglycerin ointment — The researchers will apply nitroglycerin ointment in a circular motion for 5 minutes over a 10 cm area on the anterior forearm of the chemotherapy patient.
  Arms: nitroglycerin ointment

SUMMARY:
compare the effectiveness sesame oil, aloe Vera gel, and nitroglycerin ointment prevention of phlebitis.

DETAILED DESCRIPTION:
One of the most frequent operations carried out by junior nursing professionals is peripheral intravenous cannulation. Understanding the peripheral intravenous cannulation process is crucial in light of this.

Intravenous cannulation is a challenging procedure that carries a considerable risk of complications. Pain is worsened by complications and side effects related to the cannula, such as superficial phlebitis and infiltration. If the cannulation fails or is disregarded, it might result in further treatment and transfer delays and possibly worse patient outcomes. Peripheral intravenous therapy can cause the unpleasant side effect known as chemotherapyinduced phlebitis (CIP), especially after chemotherapy. To prevent the development of (CIP), the nurses take preventative measures. The most frequent side effect of intravenous chemotherapy drug injection is vein inflammation, or phlebitis, which interferes with the treatment. Nurses have been very concerned about preventing any damage to the veins from phlebitis because they are responsible for administering chemotherapy.

Important of the study: One of the biggest health issues facing modern society is cancer. According to the World Health Organization, there is a steady upward trend in cancer incidence worldwide. Worldwide death rates from cancer are 9% due to all forms of the disease. After heart problems, cancer is the second most common cause of death in developed countries, accounting for 19% of deaths. In developing countries, cancer is the fourth most common cause of death and a contributing factor in 6% of deaths. Statistics show that over 5 million deaths worldwide are related to cancer, out of an estimated 50 million deaths annually. Chemotherapy is one of many treatment modalities used to fight cancer; it is considered a systemic approach. This method makes use of drugs that are cytotoxic. Cancer is the second leading cause of death in Iraq and the fourth leading cause in the Eastern Mediterranean region, and its incidence is rising quickly. The aging population trend, improved identification and registration, and-most importantly-increased exposure to risk factors are all contributing factors to the observed increase. Smoking is the most significant of these risk factors. Unhealthy eating habits, less exercise, other behavioral changes in lifestyle, pollution, and higher exposure to carcinogens from agriculture and industry are additional factors. With a 5.3% mortality3 rate in 2013, colorectal cancer was Iraq's ninth leading cause of death, accounting for 8341 cancerrelated deaths overall-roughly 4301 for men and 4040 for women. The National Plan of Cancer Control states that. Over the last 30 years of the 20th century, the global cancer epidemic has doubled; by 2030, it is predicted to nearly triple; and by 2050, it will increase threefold.

Chemotherapy, as a therapeutic intervention for malignancies, plays a crucial role in prolonging patients' survival rates. Nevertheless, the pharmacological agents employed in chemotherapy are associated with a myriad of deleterious side effects. Among these adverse reactions, phlebitis is a notable complication. Chemotherapy medications can harm the skin's and nails' rapidly proliferating cells. Even though some of these changes may hurt, the majority are benign and don't need medical attention. Many of them will recover after their chemotherapy course is over. Major skin changes, however, must be addressed immediately because they may result in permanent harm. small alterations to the skin When receiving chemotherapy via an IV, darker veins may appear darker and exhibit itching, dryness, redness, rashes, and peeling.

It is the most widely used way to administer chemotherapy for cancer. administered either peripherally or via central venous catheters. Absorption has greater dependability. In addition to minimizing the need for repeated injections, this route is necessary for the administration of vesicants. The risk of infection and potentially fatal sepsis is a significant side effect of intravenous (IV) chemotherapy since it allows direct access to the circulatory system.

Is the unintentional release of irritant or vesicant chemotherapy medications into the surrounding tissues at the intravenous site . A chemical that causes blisters and tissue damage is known as a vesicant. Whatever causes venous pain at the vein's location and along its length, whether or not an inflammatory response occurs us, is considered an irritant. Sloughing off of tissue, infection, pain, and impaired movement of an limb are among the possible injuries.

Using a peripheral intravenous cannula is one of a hospital nurse's most crucial responsibilities. The most common ways to get fluids into the bloods tream for chemotherapy and blood transfusions or their derivatives are intravenous therapy and fluid administration, regardless of whether the patient is being treated in an emergency room or is admitted to the hospital.4 Phlebitis occurred in as many as 70% of patients undergoing intravenous chemotherapy. Phlebitis can result in deep vein thrombosis and superficial vein thrombosis, both of which can kill and disable cancer patients. According to one study, 35-65% of cancer patients experience phlebitis brought on by chemotherapy.

Approximately 70% to 90% of patients undergoing chemotherapy will develop chemotherapyinduced phlebitis (CIP). Over half of patients die from phlebitis related to catheter use. The range of 1.3% to 61.2% represents the incidence of phlebitis. Sesame oil is important in preventing phlebitis because it can be absorbed through the skin. suggested as a preventative measure against chemotherapy-induced phlebitis. Further investigation is advised, preferably in other hospital wards and with a larger sample size.

Sesame oil application is advised as a standard hospital treatment for patients receiving chemotherapy. It is possible to conduct a similar study with a large probability sample and in a variety of settings, allowing for greater generalization of the findings. partnering with other organizations to apply cold compresses and sesame oil as a preventative measure to lower chemotherapy-associated pneumonia (CIP) in patients. Patients with cancer should learn how to recognize and report any changes in their vein health. When compared to patients who did not apply topical sesame oil on the third, fifth, or seventh day, the application of local sesame oil greatly decreased the intensity of pain on those days. It was also shown that the application of topical sesame oil sped up the recovery and healing process. The effects of topical sesame oil application on the degree of pain following chemical and boiling water burns, as well as the effects of other medicinal plants on the degree of pain and phlebitis, are proposed. Putting a compress of aloe Vera on to treat phlebitis is a novel non-pharmacological therapy approach. Aloe Vera is beneficial because it won't cause extraversion due to its low electrolyte concentrate. Aloe Vera dramatically lowered the degree of phlebitis, according to research by Anggraeni et al. An earlier study on the effects of nitroglycerin ointment on phlebitis examined the differences in incidence of angiocath-induced superficial phlebitis between clobetasol and nitroglycerin ointments. The incidence of catheter-induced phlebitis was observed to be decreased by nitroglycerin ointment, and its use was advised to avoid phlebitis in patients who require long-term5 angiocath usage. Avazeh et al. looked into the effects of topical nitroglycerine treatment on the incidence and severity of phlebitis caused by catheters. Breast cancer, which affects both men and women, is typified by the aberrant proliferation of cancerous cells in the mammary glands. Breast cancer is second in terms of overall frequency among all cancers in women, with around 1.7 million new cases identified in 2012. It is also the leading cause of cancer-related deaths among women worldwide. This accounts for roughly 12% of all newly diagnosed instances of cancer and 25% of. Globally, breast cancer is the most frequent cancer to affect women. It is the most common malignancy among Iraqis overall and accounts for almost one-third of all female cancer cases that are reported. For the past 20 years, breast cancer has been the most common malignancy among Iraqis, indicating a tendency for the disease to strike younger women. Because to early identification and effective treatment, 89% of women with breast cancer in western nations were still alive five years after receiving their diagnosis, despite the disease's high incidence rates.

The second most prevalent cause of cancer-related mortality globally and the third most common kind of cancer is colorectal cancer. Patients who have a high chance of recurrence are treated with adjuvant chemotherapy. According to GLOBOCAN 2018 data, colorectal cancer (CRC) ranks fourth in terms of diagnosis frequency and third globally in terms of fatality. The incidence of CRC varies greatly between industrialized and developing nations. CRC accounts for 6% of all cancer cases reported in Iraq.

Family history and first-degree relatives with colorectal cancer are considered high risk factors. Conversely, intermediate risk factors consist of increasing consumption of red meat, obesity, sedentary lifestyles, low consumption of fruits and vegetables, and smoking. Variations in exposure to those risk variables could lead to notable differences in cancer incidence between nations. Phlebitis in patients has been associated with the regularly used chemotherapy medication cisplatin, mostly because to its inflammatory and procoagulant characteristics. Understanding these pathways is essential to improving patient outcomes. Red blood cell procoagulant activity is increased by cisplatin treatment and is highly linked with phosphatidylserine exposure. This could contribute to the etiology of thrombophilia in breast cancer patients after treatment with cisplatin. To ensure the suppression of cancer cells that might have persisted or spread to other organs, 5- fluorouracil (5-FU) is a necessary component of systemic chemotherapy for colorectal cancer (CRC). For colorectal cancer, 5-fluorouracil (5FU) is the most frequently recommended medication. Nevertheless, recurrence after 5-FU therapy is unfortunately common and could be linked to p53-mediated WNT/β-catenin signaling, which enriches cancer stem cells in both adjuvant and palliative settings. The illness known as superficial phlebitis, which is characterized by vein inflammation, is linked to 5-fluorouracil (5-FU). Impairment of microvascular responsiveness, oxidative stress, and endothelial dysfunction are the fundamental mechanisms causing this negative effect. 5-FU causes endothelial cell injury, which raises thrombogenicity and inflammation. subsequent phlebitis, as platelet aggregation and clot formation are encouraged by the injured endothelium. This endothelial damage can 48 lead to arterial blockage because the medication increases superoxide anion levels, which lower endothelial cells' antioxidant capacity and worsen inflammation and cellular damage. One important element in the pathophysiology of vascular problems, such as phlebitis, is oxidative stress. This study's primary objective is to close this gap by comparing three methods in a clinical trial and identifying the most successful one for lowering the risk of phlebitis. among patients receiving intravenous catheter chemotherapy. Lack of proposed definitive methods for phlebitis treatment need for low-cost and novel prevention methods. Lack of comparison with other anti-phlebitis treatments. Limited discussion on potential confounding variables affecting results.

ELIGIBILITY:
Inclusion Criteria:

* adult conscious patients of both gender.
* Patients receiving chemotherapy antimetabolites (5-fluorouracil).
* Patients receiving chemotherapy alkylating agents (Cisplatin).
* Patients receiving chemotherapy through peripheral IV cannula.
* Patients breast cancer colon cancer.

Exclusion Criteria:

* Phlebitis has already appeared at the IV infusion site.
* Patients using port or central venous catheters to administer chemotherapy. - Patient radiation therapy, immunity therapy and palliative therapy
* Patients receiving chemotherapy (antitumor antibiotics, plant alkaloids).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Phlebitis Scale | 24-48 hours
  Multiple measurements will be aggregated to arrive at one reported value (phlebitis) that consists of five symptom grades were included in the chemotherapy-induced phlebitis severity scale, ranging from zero to four in severity. The National Cancer Institute Common Terminology Criteria for Adverse Events version 4 (NCI-CTCAE) (41). Which is widely used by clinical oncologists, served as the basis for the selection of grading levels. Grade zero denotes no symptoms); (grade one mild), ( grade two moderate), ( grade three marked) (and grade four severe).

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Shakhbazova A, Marsch AF. Systemic 5-fluorouracil induced lupus erythematosus: a review of the literature. Dermatol Online J. 2019 Nov 15;25(11):13030/qt3nw0p7hn. PMID 32045142
- [Result] Yousef MI, Saad AA, El-Shennawy LK. Protective effect of grape seed proanthocyanidin extract against oxidative stress induced by cisplatin in rats. Food Chem Toxicol. 2009 Jun;47(6):1176-1183. doi: 10.1016/j.fct.2009.02.007. PMID 19425235
- [Result] Kadoyama K, Miki I, Tamura T, Brown JB, Sakaeda T, Okuno Y. Adverse event profiles of 5-fluorouracil and capecitabine: data mining of the public version of the FDA Adverse Event Reporting System, AERS, and reproducibility of clinical observations. Int J Med Sci. 2012;9(1):33-9. doi: 10.7150/ijms.9.33. Epub 2011 Nov 17. PMID 22211087
- [Result] Tsimberidou AM, Braiteh F, Stewart DJ, Kurzrock R. Ultimate fate of oncology drugs approved by the us food and drug administration without a randomized Trial. J Clin Oncol. 2009 Dec 20;27(36):6243-50. doi: 10.1200/JCO.2009.23.6018. Epub 2009 Oct 13. PMID 19826112
- [Result] Sudhakar S, Jacob A, Hegde NN, Chaudhary RK, Mateti UV, Shetty V. Evaluation of chemotherapy infusion and phlebitis among cancer patients: A prospective observational single-center study. J Oncol Pharm Pract. 2023 Dec;29(8):1944-1950. doi: 10.1177/10781552231161517. Epub 2023 Mar 5. PMID 36872649
- [Result] Outcomes of Patients with Chronic Lymphocytic Leukemia Treated with Chemotherapy in Middle Euphrates Region of Iraq: Data from Developing CountryMjali A. 2020;12
- [Result] Johnson CM, Wei C, Ensor JE, Smolenski DJ, Amos CI, Levin B, Berry DA. Meta-analyses of colorectal cancer risk factors. Cancer Causes Control. 2013 Jun;24(6):1207-22. doi: 10.1007/s10552-013-0201-5. Epub 2013 Apr 6. PMID 23563998
- [Result] Some Facts About Cancers in Karbala province of Iraq, 2012-2020Mjali A, Baroodi B. Asian Pacific Journal of Cancer Care.2020;5.
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Argiles G, Tabernero J, Labianca R, Hochhauser D, Salazar R, Iveson T, Laurent-Puig P, Quirke P, Yoshino T, Taieb J, Martinelli E, Arnold D; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Localised colon cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2020 Oct;31(10):1291-1305. doi: 10.1016/j.annonc.2020.06.022. Epub 2020 Jul 20. No abstract available. PMID 32702383
- [Result] Iraqi Cancer Board: Results of the Iraqi Cancer Registry 2011. Baghdad, Iraqi Cancer Registry Center: Ministry of Health, 2013.
- [Result] Alwan NA. Breast cancer: demographic characteristics and clinico-pathological presentation of patients in Iraq. East Mediterr Health J. 2010 Nov;16(11):1159-64. PMID 21218740
- [Result] International Agency for Cancer Research (IARC); World health Organization: GLOBOCAN 2012 v1.1, Cancer Incidence and Mortality Worldwide: IARC Cancer Base, 2012, No. 11 [Online], Available from: http://globocan.iarc.fr , accessed on 16/05/2016.
- [Result] American Cancer society (A): Breast cancer:Facts and Figures 2015-2016. Atlanta:Author, 2016, [Online], Available from: www.cancer.org/cancerfactsstatistics/acspc-046381 , accessed on 26/01/2016.
- [Result] Akbari H, Raufi S, Hekmat po D , Anbari K (2014). Comparaing the effect of Nitroglycerin and Clobetazol Ointments on Prevention of Superficial Intravenous Catheter Induced Phlebitis. Evide Based Care, 4, 71-80
- [Result] Annai S, Deepa R. Effectiveness of aloe vera gel application on phlebitis. Nurse Care Open Acces J. 2023;9(3):122-128. DOI: 10.15406/ncoaj.2023.09.00271
- [Result] Mohammadyan S, Seidi J, Nouri B, Fathi M. [A Comparative Study on the Effect of Aloe Vera and Nitroglycerin Ointment on the Incidence and Severity of Phlebitis Caused by the Peripheral Catheter]. Sci J Kurdistan Univ Med Sci. 2020;25(2):44-53. Persian
- [Result] Ghazanfari Z, Foroghamari G, Mirhosseini M. [The nursing staff view about barriers of using pain relief methods]. Crit Care Nurs. 2011;3(4):153-6. Persian
- [Result] Dorchin M, Dorchin A, Attar N, Moradi N, Sharifzadeh Z (2021) The Role of Rubbing Sesame Oil in Improving Chemotherapy Induced Phlebitis in Cancer Patients at Raha Cancer Clinic: Dezful. J Pharma Care Health Sys. 8:234.
- [Result] Behnamfar N, Parsa Yekta Z, Mojab F, Kazem Naeini SM. The effect of nigella sativa oil on the prevention of phlebitis induced by chemotherapy: a clinical trial. Biomedicine (Taipei). 2019 Sep;9(3):20. doi: 10.1051/bmdcn/2019090320. Epub 2019 Aug 27. PMID 31453801
- [Result] Shafipour SZ, Mosayebi N, Asgari F, Atrkarroushan Z , Pasdaran A (2017). Effect of External Use of Sesame Oil in the Prevention of Chemotherapy-Induced Phlebitis in Children
- [Result] Gonzalez Lopez JL, Arribi Vilela A, Fernandez del Palacio E, Olivares Corral J, Benedicto Marti C, Herrera Portal P. Indwell times, complications and costs of open vs closed safety peripheral intravenous catheters: a randomized study. J Hosp Infect. 2014 Feb;86(2):117-26. doi: 10.1016/j.jhin.2013.10.008. Epub 2013 Dec 1. PMID 24373830
- [Result] Y. Gao, T. Jiang, S. Mei, S. Zhang, C. Zhu, Y. Sun. Meta-analysis of Aloe vera for the prevention and treatment of chemotherapy-induced phlebitis. Int J Clin Exp Med. 9(6); 2016: 9642- 50
- [Result] Kaewwilai, S., & Uadrang, S. (2022). อุบัติ การณ์ การ เกิด หลอดเลือด ด า อักเสบ อุด ตัน ใน ผู้ ป่ วย มะเร็ง ที่ ได้ รับ ยา เคมี บ าบัด. Journal of The Department of Medical Services, 47(3), 27-31
- [Result] Ahmed, K. A., & Hamawandi, N. M. Assessment of peripheral intravenous cannula insertion pr actice among health care workers of sulaimani surgical teaching hospital, sulaimani, iraq
- [Result] Gonzalez T. Chemotherapy extravasations: prevention, identification, management, and documentation. Clin J Oncol Nurs. 2013 Feb;17(1):61-6. doi: 10.1188/13.CJON.61-66. PMID 23372097
- [Result] Patrick, C. N. (2010). Diagnosis and Treatment, 82(2). https://doi.org/10.1016/S0195- 5616(00)06007-1.
- [Result] Hayder, A. J., & Mohammed, S. J. (2018). Effectiveness of an Education Program on Nurses' Knowledge Concerning Side Effect of Chemotherapy in Baghdad Teaching Hospitals. Indian Journal of Public Health Research & Development, 9(8).
- [Result] Harris V, Hughes M, Roberts R, Dolan G, Williams EM. The Development and Testing of a Chemotherapy-Induced Phlebitis Severity (CIPS) Scale for Patients Receiving Anthracycline Chemotherapy for Breast Cancer. J Clin Med. 2020 Mar 5;9(3):701. doi: 10.3390/jcm9030701. PMID 32150833
- [Result] National Cancer Control Plan of Egypt, (2020). http:// ahfonline. net/ files/ mp/ Cancer %20Control %20Plan.pdf
- [Result] MO) Ministry of Health. (2013). Iraqi Cancer Registry Center, Baghdad
- [Result] Mimoz O, Villeminey S, Ragot S, Dahyot-Fizelier C, Laksiri L, Petitpas F, Debaene B. Chlorhexidine-based antiseptic solution vs alcohol-based povidone-iodine for central venous catheter care. Arch Intern Med. 2007 Oct 22;167(19):2066-72. doi: 10.1001/archinte.167.19.2066. PMID 17954800
- [Result] Ali HD. Quality of life and its related factors in cancer patients undergoing chemotherapy. J Kerm University Med Sci. 2006; 1(2): 119-110.
- [Result] Otto SE. Oncology Nursing. Ed. 4th ed Mosby, Toronto. Harcourt Health Sciences CO. 2001
- [Result] Shojaei Tehrani Hossein. Textbook of Medicine, Prevention and Social. Chronic NonCommunicable Diseases and Common Infectious Diseases. Med Sci Tehran. 2003;4(1): 28-25.
- [Result] El-Sayad, H. E., Aboalizm, S. E., & Abd Elhy, A. H. (2023). Effect of preventive measures on chemotherapy induced phlebitis among patients with cancer. Menoufia Nursing Journal, 8(1), 187-202.
- [Result] Hussin, B. K. (2021 Prevention of Extravasation Non-Cytotoxic Agents (Review Study). Himalayan Journal of Nursing and Midwifery, 1(5).
- [Result] Carr PJ, Glynn RW, Dineen B, Kropmans TJ. A pilot intravenous cannulation team: an Irish perspective. Br J Nurs. 2010 May 27-Jun 9;19(10):S19-27. doi: 10.12968/bjon.2010.19.Sup3.48214. PMID 20622770
- [Result] Carr PJ, Glynn RW, Dineen B, Devitt D, Flaherty G, Kropmans TJ, Kerin M. Interns' attitudes to IV cannulation: a KAP study. Br J Nurs. 2011 Feb 24-Mar 9;20(4):S15-20. doi: 10.12968/bjon.2011.20.4.S15. PMID 21471870